CLINICAL TRIAL: NCT05143723
Title: Luteal Phase Support With Daily Administration of Gonadotropin-releasing Hormone Agonist Compared to Progesterone/Estradiol in IVF/ICSI Cycles With Ovulation Triggering With GnRH-a
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuban State Medical University (Other)
Responsible Party: Principal Investigator, Alisa Baklakova, doctor gynecologist, Kuban State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04081990
Record Dates: First submitted 2021-11-07; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- agonist group (Experimental): Patients of the first group received GNRH-a for LPS at a dose of 0.2 mg, subdermally, daily from the second day after TVOP till 8 weeks of pregnancy.
  Interventions: Drug: Gonadotropin-releasing hormone agonist
- group of progesterone and estradiol (Active Comparator): The second group of patients received progesterone as LPS at a dosage of 30 mg per day, per os, and estradiol at a dosage of 3 mg per day, transdermally starting from the second day after TVOP till 8 weeks of pregnancy
  Interventions: Drug: Gonadotropin-releasing hormone agonist

INTERVENTIONS:
Drug: Gonadotropin-releasing hormone agonist — luteal phase support with gonadotropin-releasing hormone agonist

SUMMARY:
Purpose: To determine the efficacy and safety of daily injections of gonadotropin-releasing hormone agonist in comparison with the standard strategy of supporting the luteal phase in protocols with gonadotropin-releasing hormone antagonists, in patients at risk of developing ovarian hyperstimulation syndrome and changing the trigger to a gonadotropin-releasing hormone agonist.

Materials and Methods: This prospective, controlled, randomized study, conducted at the Clinic of the Federal State Budgetary Educational Institution of Higher Education of the KubSMU of the Ministry of Health of Russia, included 102 patients at risk of developing ovarian hyperstimulation syndrome, who were on protocols with gonadotropin-releasing hormone antagonists and changing the ovulation trigger to a gonadotropin-releasing hormone agonist. All patients underwent blastocyst transfer on day 5. Patients of the first group (n = 51) received as support for the luteal phase gonadotropin-releasing hormone agonist daily 0.2 mg, subdermally, patients of the second group (n = 51) progesterone 10 mg 3 times a day, orally and estradiol 1 mg 3 times a day, transdermal. The level of progesterone on the day of transfer, the incidence of clinical pregnancy, and the incidence of ovarian hyperstimulation syndrome in both groups were compared.

DETAILED DESCRIPTION:
This prospective randomized study was conducted at the Clinic of the Federal State Budgetary Educational Institution of Higher Education of the Kuban State Medical University of the Ministry of Health of Russia from January 2020 till April 2021 and was approved by the ethical committee of the FSBEI HE KubSMU of the Ministry of Health of Russia Protocol No. 83 dated 07.11.2019. It included 102 patients at risk of developing OHSS, all of whom gave written informed voluntary consent. Inclusion criteria were: age - from 20 to 40; AMH - more than 2.5 ng/ml; the number of antral follicles (AFC) - more than 15 (menstrual cycle days 1-5); stimulation of ovarian function in the protocol with GnRH-antagonist in IVF/ICSI cycles, with the change of the ovulation trigger to GnRH-a; tubal, unspecified and anovulatory infertility; body mass index (BMI) from 18 to 29 (inclusive); 15 or more follicles per day of ovulation trigger injection.

Exclusion criteria: presence of external genital endometriosis; male factor of infertility; hydrosalpinx and/or tubo-ovarian formation (on one or both sides) according to hysterosalpingography and/or ultrasound investigation; malformations of internal genital organs, including conditions after surgical correction of malformations of internal genital organs; acquired deformities of the uterine cavity, in which embryo implantation or pregnancy is impossible; contraindications to the IVF/ICSI program; severe systemic diseases; cycles with cryopreserved sperm or oocytes; oocyte donation. The patients were divided into two groups using the envelope method. On days 2-5 of the menstrual cycle, a study of the level of blood hormones was carried out: follicle-stimulating hormone (FSH), luteinizing hormone (LH), progesterone, and estradiol, as well as transvaginal ultrasonography of the pelvic organs to determine the number of antral follicles (AFC) and exclusion of contraindications for the start of COS. Then СOS was carried out using gonadotropins, menotropins. The standard daily starting dose of stimulant drugs was determined according to age, BMI, original FSH, AFC, and ovarian response in women undergoing previous IVF/ICSI cycles. The ovarian response was assessed using folliculometry, starting from 5-6 days of COS, when two follicles with an average diameter of more than 14 mm or one more than 16 mm were reached, GnRH-ant was prescribed at a dose of 0.25 mg daily. Ovulation trigger (GnRH-a) was introduced on condition that two or more follicles with a diameter of 17-18 mm were reached; after 36 hours, transvaginal ovarian puncture (TVOP) was performed under ultrasound control. All mature eggs (ova) were fertilized using IVF or ICSI methods. Fertilization was assessed after about 20 hours, and the embryos were transferred into the uterine cavity on day 3 or 5. LPS in all patients started the day after oocyte retrieval and continued until 8 weeks of gestation in case of positive result.

Patients of the first group (n=51) received GNRH-a for LPS at a dose of 0.2 mg, subdermally, daily from the second day after TVOP. The second group of patients (n=51) received progesterone as LPS at a dosage of 30 mg per day, per os, and estradiol at a dosage of 3 mg per day, transdermally starting from the second day after TVOP till 8 weeks of pregnancy. The embryo transfer was carried out 3-5 days after TVOP, one or two embryos were transferred, depending on the morphological assessment of the embryo. On the day of transfer, a study of the level of progesterone in the peripheral blood was carried out. Pregnancy testing was performed by determining the level of β-hCG in the peripheral blood 14 days after the embryo transfer. Data were collected on participant characteristics, COS, and embryology. Characteristics included: patient's age, characteristics of ovarian reserve (AMH, FSH), type, duration and cause of infertility, duration of COS, the total dose of gonadotropin treatment, endometrial thickness on the day of ovulation trigger administration, number of oocytes and embryos retrieved. The outcomes were positive dynamics of β-hCG growth and clinical indicators of pregnancy. Clinical pregnancy was defined as an ongoing pregnancy with ultrasound imaging of the ovum and fetal heart rate.

Statistical analysis of data was carried out using STATISCA 10 package (Tibco, USA). Spearman's rank correlation coefficient, Mann-Whitney U test, Pearson's Chi-square test, Maximum likelihood Chi-square tests were used. p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age - from 20 to 40; AMH - more than 2.5 ng/ml
* Number of antral follicles (AFC) - more than 15 (menstrual cycle days 1-5)
* Stimulation of ovarian function in the protocol with GnRH-ant in IVF/ICSI cycles, with the change of the ovulation trigger to GnRH-a
* Tubal, unspecified and anovulatory infertility
* Body mass index (BMI) from 18 to 29 (inclusive)
* 15 or more follicles per day of ovulation trigger injection

Exclusion Criteria:

* Presence of external genital endometriosis
* Male factor of infertility
* Hydrosalpinx and/or tubo-ovarian formation (on one or both sides) according to hysterosalpingography and/or ultrasound investigation
* Malformations of internal genital organs, including conditions after surgical correction of malformations of internal genital organs
* Acquired deformities of the uterine cavity, in which embryo implantation or pregnancy is impossible
* Contraindications to the IVF/ICSI program; severe systemic diseases
* Cycles with GnRH antagonists

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate and clinical pregnancy rate | 35 day after embryo transfer
  Pregnancy was assessed by measuring serum β-hCG levels 14 days after embryo transfer, and clinical pregnancy was confirmed by the presence of an intrauterine gestational sac on ultrasound examination 5 weeks after embryo transfer. Clinical pregnancy rate was calculated as the number of clinical pregnancies divided by the number of embryo transfer procedures

SECONDARY OUTCOMES:
serum progesterone level | Day 5 after embryo transfer
  A study of the level of progesterone in the blood serum was carried out on the day of transfer of emryos

CONTACTS AND LOCATIONS:
Locations (1):
- Alisa Baklakova, Krasnodar, Krasnodarskiy Kray, Russia

IPD SHARING:
Plan to Share IPD: Undecided